CLINICAL TRIAL: NCT05500781
Title: Coaching HER: Eliminating Gender Stereotypes in Sport Coaching
Brief Title: Online Program for Coaching Girls: Coaching HER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Unilever R&D (Industry); Nike (Industry); Laureus (Unknown); University of West England (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY00015642
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Intervention; Waitlist Control
Keywords: Athletes; Girls; Coaches; Web-based; Coach Education; Gender Stereotypes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coaching HER (Experimental): Participants in the interventional condition will take part in an online program consisting of 6 modules over 2 weeks
  Interventions: Behavioral: Coaching HER
- Waitlist Control (No Intervention): Participants will not be explicitly told their study condition, although they will be made aware of the assessment time points and whether they receive the intervention between T1 and T2 (intervention) or after T2 (waitlist control). Following completion of post-intervention assessments (T2), the control condition will participate in the intervention; but, they will not be monitored or assessed.

INTERVENTIONS:
Behavioral: Coaching HER — The CoachingHER coach education program is a six-module online program aimed at upskilling coaches in [the effectiveness, feasibility, and acceptability of the Coaching HER; the first online program aimed at reducing gender stereotypes for coaches]. Each module will take approximately 20 minutes to complete and consists of educational content, interactive elements (quizzes, checklists, opinion polls, reflective exercises), and additional resources.
  Arms: Coaching HER

SUMMARY:
Despite the numerous physical and psychological benefits of taking part in sport, studies consistently show that only 15% of adolescent girls globally meet the recommended daily exercise guidelines (Guthold et al., 2018). The team climate, created by coaches, has been identified as a critical factor in both girls' participation in, and enjoyment of, sport and movement (CITE). Research indicates that girls disengage from sport because of body image concerns, uncomfortable and objectifying uniforms, appearance-related teasing from peers and coaches, untrained coaches, and negative team cultures (Murray et al., 2021; Vani et al., 2021).

help coaching girls books as another form of media that produces "commonsense proof" of girls' sport inferiority, essentializes gender differences, reifies the gender binary (Kane, 1995), and marginalizes the sport participation of girls.

The beliefs, values and expectations of significant adults can positively or negatively influence self-perceptions, motivation, experiences, and behaviors of children (Fredricks & Eccles, 2005; Brustad et al., 2001) and also directly influence the coaching behaviors of adults (Cassidy et al., 2005).

The 'coaching girls' books examined for this study were formulaic products written from a perspective of difference, "despite extensive evidence from meta-analysis research of gender differences which supports the gender similarity hypothesis" (Hyde, 2005, p.590).

ambivalent and primarily non-research based messages contained within the books trivialize, misrepresent, distort, and marginalize girls' emotions, thoughts, relationships, skills and behaviors in sport contexts (Birrell & Theberge, 1994), while upholding coaching boys as normative praxis. Coaching girls books appear to "help" coaches of female athletes, while simultaneously reifying gender stereotypes that undermine female empowerment that can occur in and through sports.

Praxis based on gendered beliefs of inherent difference is dangerous as it can undermine male-female relationships as well as beliefs of equality, and deprive all children of the opportunity to develop their full human potential (Barnett & Rivers, 2004). Coaches must be aware that coaching is a gendered practice in which beliefs and values are enacted, sometimes in ways that limit the experiences of their athletes.

On the other hand, sport participation can improve girls' self perceptions and lead to accrual of health and development assets if the coach and adults in the context are aware of the gendered nature of sport, and strive to eliminate deleterious effects (LaVoi, 2018).

This study will test an educational program for coaches aimed at reducing gender essentialist beliefs and gender stereotypes of coaches, to improve the sport experience for girls.

ELIGIBILITY:
Inclusion Criteria:

* Current Coaches of adolescent girls
* English speaking
* U.S. resident

Exclusion Criteria:

* Participants under 18 years of age
* Coaches outside of the US
* Coaches who only coach adult women or men/boys

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Change in coaches' self-efficacy in tackling gender stereotypes | Baseline, pre-intervention; immediately after the intervention (2 weeks later)
  Change in coaches' self-efficacy in tackling gender stereotypes assessed via the Coach Confidence: Gender Stereotypes In Sport (modified from Vaughan et al., 2004)

SECONDARY OUTCOMES:
Change in coaches' self-efficacy in tackling gender essentialist beliefs | Baseline, pre-intervention; immediately after the intervention (2 weeks later)
  Process Outcome
Total feasibility, acceptability, and adherence of the intervention (assessed via a self-report questionnaire) | Immediately after the intervention
  Assess the feasibility, acceptability, and adherence of the CoachingHER coach education program

OTHER OUTCOMES:
Total acceptability of the intervention (assessed via a self-report questionnaire) | Immediately after the intervention
  Coaches will complete feasibility and acceptability measures via a self-report questionnaire on a scale from 1 (Strongly Disagree) to 5 (Strongly Agree) within the following domains: 1) affective attitude (e.g., I liked this program); 2) burden (e.g., it was easy to follow the content of the program; 3) ethicality (e.g., I think this program is appropriate for coaches in my sport; 4) self-efficacy (e.g., I am confident that I will use the techniques I learned from this program); 5) perceived effectiveness (e.g., the program was successful in improving my knowledge about gender stereotypes); and 6) content (e.g., how easy or difficult was it to follow the program?).
Total intervention adherence (assessed through session completion) | Immediately after the intervention
  Total intervention adherence will be assessed by the investigators as number of participants who complete the full intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnett, R., & Rivers, C. (2004). Same difference: How gender myths are hurting our relationships, our children, and our jobs. New York: Basic Books.
- [Background] Birrell, S., & Theberge, N. (1994). Ideological control of women in sport. In D.M. Costa & S.R. Guthrie (Eds.), Women and sport: Interdisciplinary perspectives (pp. 341-359). Champaign, IL: Human Kinetics
- [Background] Brustad, R.J., Babkes, M.L., Smith (2001). Youth in sport: Psychological considerations (2nd ed.). New York: John Wiley & Sons
- [Background] Cassidy, T., Jones, R., & Potrac, P. (2005). Understanding sports coaching: The social, cultural and pedagogical foundations of coaching practice. New York: Routledge.
- [Background] Fredricks, J.A, & Eccles, J.S. (2005). Family socialization, gender, and sport motivation and involvement. Journal of Sport & Exercise Psychology, 27, 3-31. https://doi.org/10.1123/jsep.27.1.3
- [Background] Guthold R, Stevens GA, Riley LM, Bull FC. Worldwide trends in insufficient physical activity from 2001 to 2016: a pooled analysis of 358 population-based surveys with 1.9 million participants. Lancet Glob Health. 2018 Oct;6(10):e1077-e1086. doi: 10.1016/S2214-109X(18)30357-7. Epub 2018 Sep 4. PMID 30193830
- [Background] Hyde JS. The gender similarities hypothesis. Am Psychol. 2005 Sep;60(6):581-592. doi: 10.1037/0003-066X.60.6.581. PMID 16173891
- [Background] Kane, M. J. (1995). Resistance/transformation of the oppositional binary: Exposing sport as a continuum. Journal of Sport and Social Issues, 19(2), 191-218. https://doi.org/10.1177/019372395019002006
- [Background] LaVoi, N.M. (2018). Girls' physical activity participation: A best practices model and summary. In N.M. LaVoi (Ed.) The 2018 Tucker Center research report, developing physically active girls: An evidence-based multidisciplinary approach (pp. 197-213). Minneapolis, MN
- [Background] Murray, R. M., Sabiston, C. M., Coffee, P., & Kowalski, K. C. (2021). Strengthening the relationship between physical activity and physical self-concept: The moderating effect of controllable attributions. Psychology of Sport and Exercise, 52, 101828.
- [Background] Vani, M. F., Murray, R. M., & Sabiston, C. M. (2021). Body image and physical activity. Essentials of exercise and sport psychology: An open access textbook, 150-175.